CLINICAL TRIAL: NCT06848309
Title: Dissecting Human Immune Responses to Infection with Influenza or SARS-CoV-2
Acronym: WU 437
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Mudd, Principal Investigator, Washington University School of Medicine
Other Study IDs: 202411171; U19AI181103 (NIH)
Record Dates: First submitted 2025-02-12; First posted 2025-02-27 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Influenza; SARS-CoV-2 (COVID-19) Infection; Immune Response of Host
Keywords: influenza vaccines; COVID-19 vaccines; bronchoscopy; nasopharyngeal sampling; saliva
MeSH Terms: conditions — Influenza, Human; COVID-19; Infections | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, nasopharyngeal swabs, saliva, bronchoalveolar lavage fluid, endobronchial biopsy tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Uninfected Cohort: Subjects that have received an FDA-approved seasonal influenza and/or SARS-CoV-2 vaccine within the past 12 months and not experienced a documented influenza or SARS-CoV-2 infection since receiving the vaccine dose.
  Interventions: Procedure: Bronchoscopy
- Seasonal Influenza Infected, Not Recently Vaccinated Cohort: CLIA-approved influenza test positive in participants with an acute illness and active symptoms of a respiratory viral infection that triggered the clinical testing. Participants in this group have not received a seasonal influenza vaccine within the last 12 months.
  Interventions: Procedure: Bronchoscopy
- Seasonal Influenza Infected, Recently Vaccinated Cohort: CLIA-approved influenza test positive in participants with an acute illness and active symptoms of a respiratory viral infection that triggered the clinical testing. Participants in this group received a seasonal influenza vaccine within the last 12 months.
  Interventions: Procedure: Bronchoscopy
- SARS-CoV-2 Infected, Not Recently Vaccinated Cohort: CLIA-approved SARS-CoV-2 test positive in participants with an acute illness and active symptoms of a respiratory viral infection that triggered the clinical testing. Participants in this group have not received a COVID-19 vaccine within the last 12 months.
  Interventions: Procedure: Bronchoscopy
- SARS-CoV-2 Infected, Recently Vaccinated Cohort: CLIA-approved SARS-CoV-2 test positive in participants with an acute illness and active symptoms of a respiratory viral infection that triggered the clinical testing. Participants in this group received a COVID-19 vaccine within the last 12 months.
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Some participants in all 5 groups may undergo an optional bronchoscopy procedure with bronchoalveolar lavage and endobronchial biopsy collection if they choose.

SUMMARY:
The purpose of this study is to evaluate the virus-specific immune response in people who are symptomatic with confirmed influenza or COVID-19. We will study the immune response of people who have and who have not been vaccinated with the seasonal influenza and COVID-19 vaccines within the past year. All participants will have data collected and blood, saliva, and nasal swabs performed at five separate visits; 1) at study enrollment, 2) on study day 7, 3) on or between study days 10 to 28, 4) on study day 90, and 5) on study day 180. For participants who agree to the optional sub-study, bronchoscopy with bronchoalveolar lavage (BAL) and endobronchial biopsy (EBBx) will be performed once between study days 10 and 28 and once at study day 180. As part of the bronchoscopy procedure, two chest x-rays will be performed. The bronchoscopy and chest x-ray procedures are not required for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have presented with acute, symptomatic seasonal influenza or SARS-CoV-2 infection proven by an approved CLIA certified test and be enrolled in study while still symptomatic or within 72 hours of the resolution of viral respiratory illness symptoms.
* Alternatively, uninfected participants in the control cohort must have received an FDA-approved seasonal influenza and/or SARS-CoV-2 vaccine within the past 12 months and not experienced a documented influenza or SARS-CoV-2 infection since receiving that most recent vaccine dose.
* Participants must be able to understand and provide full written informed consent.
* Participants must be male or female between the ages of 18 and 60.
* Participants must be in stable health, as determined by medical history and targeted physical exam related to that history.

Exclusion Criteria:

* Co-infection with any respiratory virus in addition to the index influenza or SARS-CoV-2 infection on a multi-plex viral testing panel.
* Severe illness with anticipated need for hospitalization for the index infection.
* Current or previous diagnosis of an immunocompromising condition.
* Receipt of systemic immunosuppressants or immune-modifying drugs for > 14 days in total within 6 months prior to screening or is anticipating the need for immunosuppressive treatment at any time during study participation.
* Current symptomatic acute or unstable chronic disease requiring medical or surgical care, to include significant change in therapy or hospitalization, at the discretion of the investigator. Any known diagnosed chronic pulmonary, cardiovascular, renal, hepatic, hematologic, or metabolic disorder with the exception of isolated treated hypertension.
* Known chronic neurologic or neurodevelopmental condition including spinal cord injury with resultant weakness of any kind (this does not exclude patients with chronic back pain or previous disk herniation/back surgery, only patients with documented weakness, quadriplegia or paraplegia). This exclusion criterion does not exclude from the study individuals with recurrent migraine headaches as their only chronic neurologic condition.
* Active cancer diagnosis, including any cancer that has not been in remission for at least 1 year. Isolated basal or squamous cell skin cancers are not excluded.
* History of excessive alcohol consumption, drug abuse, psychiatric conditions, social conditions, or occupational conditions that in the opinion of the investigator would preclude compliance with the study.
* Body Mass Index (BMI) > 40
* Pregnant women and nursing mothers or women who are planning to become pregnant during the study interval.
* Have donated blood, blood products or bone marrow within 30 days before study entry or plan to donate blood at any time during the duration of study participation or up to 30 days after the last study blood draw.
* Current ongoing participation in a clinical trial evaluating an investigational agent, unless the trial is in follow-up only and the last dose of the investigational agent was taken > 30 days or > 5 half-lives prior to enrollment, whichever is greater.
* Any condition in the opinion of the investigator that would interfere with the safe and proper conduct of the study.

For participants willing to undergo bronchoscopy:

* Coagulopathy as defined by screening safety labs that reveal an INR > 1.4, at PTT > 40, or a platelet count < 100,000 precludes participation in the bronchoscopy procedure.
* Evidence of ongoing significant pulmonary disease on the day of bronchoscopy, including pulse oximetry with oxygen saturation of 92% or less on room air, or infiltrate or pleural effusion noted on an upright PA and lateral chest x-ray performed on the day of bronchoscopy.
* Allergy or contraindication to anesthesia for participants willing to undergo bronchoscopy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is healthy, non-pregnant or breastfeeding adults ages 18-60 with recent vaccination against seasonal influenza and/or SARS-CoV-2 or with acute seasonal influenza infection or acute SARS-CoV-2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
To measure the difference in the concentration of systemic and mucosal influenza-specific or SARS-CoV-2-specific IgG and IgA in the blood, saliva, nasopharynx, and lower airways and how these concentrations change over time following acute infection | At study enrollment (day 0) which will occur during active symptomatic viral infection and at 6 months after study enrollment

SECONDARY OUTCOMES:
To measure the difference between the systemic and mucosal influenza- and SARS-CoV-2-specific IgG and IgA antibody concentration in patients who received and those who did not receive a seasonal vaccine in the past 12 months | At study enrollment (day 0) which will occur during active symptomatic viral infection and at 6 months after study enrollment
To measure the frequency of influenza- and SARS-CoV-2-specific CD4+ and CD8+ T cells in the blood, nasopharynx, lower airways, and lung tissue in individuals who received and those that did not receive the seasonal vaccine in the previous 12 months | At study enrollment (day 0) which will occur during active symptomatic viral infection and at 6 months after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Mudd, MD, PhD, Principal Investigator — Washington University in Saint Louis School of Medicine
Locations (1):
- Washington University in Saint Louis Department of Emergency Medicine, Emergency Care Research Core, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Completely de-identified individual participant-level data will be provided to the scientific community following study completion and publication through reasonable request of the study principal investigator via email.
Supporting Information: Study Protocol, ICF
Time Frame: IPD and supporting information will be available on the date of study results publication and will be made available for 10 years following publication of study results.
Access Criteria: Researchers performing secondary analyses of study results may request any generated deidentified individual participant level data following data or material transfer agreement completion.